CLINICAL TRIAL: NCT03980990
Title: Metformin Continuation Versus Interruption Following Coronary Angiography: a Pilot Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jay Shavadia, Assistant Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OA-UofS-778
Record Dates: First submitted 2019-06-05; First posted 2019-06-10 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Acute Coronary Syndrome; Unstable Angina; Diabetes Mellitus; Metformin Adverse Reaction
Keywords: metformin; diabetes; pci; percutaneous coronary intervention; unstable angina; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metformin Continuation (Experimental): Patients undergoing angiography will continue their metformin without interruption at their next scheduled dose following angiography.
  Interventions: Drug: Metformin
- Metformin Interruption (No Intervention): Patients undergoing angiography will interrupt their metformin for 48 hours post angiography.

INTERVENTIONS:
Drug: Metformin — Continuation of Metformin
  Arms: Metformin Continuation

SUMMARY:
This pilot randomized controlled trial aims to evaluate the feasibility for safety examination of continued metformin therapy in patients with type 2 diabetes (T2D) following invasive coronary angiography. Metformin will be continued until coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. On metformin therapy
3. Angiography for ACS or elective non-ACS related indications
4. Informed consent received

Exclusion Criteria:

1. Cardiogenic shock prior to randomization
2. Cardiac arrest prior to randomization
3. Established severe CKD (eGFR<30, or on dialysis)
4. Chronic liver disease
5. Need for CABG within 48 hours of hospitalization
6. Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk if the investigational therapy is initiated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-06-17 (Estimated); Study Completion 2020-06-17 (Estimated)

PRIMARY OUTCOMES:
Lactic Acidosis | 48-72 hours (or 72 hours for patients with staged PCI procedures within 48 hours of randomization)
  Lactate Level >5 mmol/L and HCO3<18

SECONDARY OUTCOMES:
Acute Kidney Injury | 48-72 hours (or 72 hours for patients with staged PCI procedures within 48 hours of randomization)
  Rise in baseline creatinine >/= 25% or 27 umol/L
All cause mortality at hospital discharge | Duration of hospital admission
  Death in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jay Shavadia, MD, Principal Investigator — University of Saskatchewan, Department of Medicine, Division of Cardiology
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salpeter SR, Greyber E, Pasternak GA, Salpeter EE. Risk of fatal and nonfatal lactic acidosis with metformin use in type 2 diabetes mellitus. Cochrane Database Syst Rev. 2010 Apr 14;2010(4):CD002967. doi: 10.1002/14651858.CD002967.pub4. PMID 20393934
- [Background] Misbin RI, Green L, Stadel BV, Gueriguian JL, Gubbi A, Fleming GA. Lactic acidosis in patients with diabetes treated with metformin. N Engl J Med. 1998 Jan 22;338(4):265-6. doi: 10.1056/NEJM199801223380415. No abstract available. PMID 9441244
- [Background] Oktay V, Calpar Cirali I, Sinan UY, Yildiz A, Ersanli MK. Impact of continuation of metformin prior to elective coronary angiography on acute contrast nephropathy in patients with normal or mildly impaired renal functions. Anatol J Cardiol. 2017 Nov;18(5):334-339. doi: 10.14744/AnatolJCardiol.2017.7836. Epub 2017 Oct 31. PMID 29111980
- [Background] Zeller M, Labalette-Bart M, Juliard JM, Potier L, Feldman LJ, Steg PG, Cottin Y, Roussel R. Metformin and contrast-induced acute kidney injury in diabetic patients treated with primary percutaneous coronary intervention for ST segment elevation myocardial infarction: Amulticenter study. Int J Cardiol. 2016 Oct 1;220:137-42. doi: 10.1016/j.ijcard.2016.06.076. Epub 2016 Jun 23. PMID 27376570
- [Background] Maznyczka A, Myat A, Gershlick A. Discontinuation of metformin in the setting of coronary angiography: clinical uncertainty amongst physicians reflecting a poor evidence base. EuroIntervention. 2012 Jan;7(9):1103-10. doi: 10.4244/EIJV7I9A175. PMID 21959259